CLINICAL TRIAL: NCT07361705
Title: An Open-Label, Multicentre, Phase 1 Clinical Study to Evaluate the Safety and Efficacy of Zorifertinib Combined With Osimertinib in Patients With Advanced Non-Small Cell Lung Cancer With Meningeal Progression After Osimertinib Treatment
Brief Title: Zorifertinib With Osimertinib for NSCLC With Meningeal Progression
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alpha Biopharma (Jiangsu) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AZD3759-005
Record Dates: First submitted 2025-12-04; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Patients With Advanced Non-small Cell Lung Cancer With Meningeal Progression After Osimertinib Treatment
Keywords: NSCLC; Leptomeningeal Metastases; Leptomeningeal Carcinomatosis; Meningeal Metastases; EGFR; Osimertinib, Zorifertinib
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — AZD3759; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zorifertinib + Osimertinib (Dose Escalation) (Experimental): All enrolled participants will receive the investigational combination therapy of Zorifertinib and Osimertinib. This is a Phase 1 study consisting of a dose escalation part (Part A) and a dose expansion part (Part B). In Part A, Zorifertinib dose will be escalated (starting at 100 mg twice daily) alongside a fixed dose of Osimertinib (80 mg once daily) using a "3+3" design to determine the recommended dose. In Part B, additional participants will receive the combination at the recommended dose to further evaluate safety, efficacy, and pharmacokinetics. Treatment continues until disease progression, unacceptable toxicity, or meeting other discontinuation criteria.
  Interventions: Drug: Zorifertinib and Osimertinib Combination Therapy

INTERVENTIONS:
Drug: Zorifertinib and Osimertinib Combination Therapy — Zorifertinib is an oral tablet (50 mg or 100 mg). Osimertinib is an oral tablet (80 mg). In this Phase 1 study, all participants will receive the combination. Osimertinib is given at a fixed dose of 80 mg once daily. Zorifertinib is given twice daily, with dose levels under evaluation (starting at 100 mg BID, potentially escalating to 150 mg BID, 200 mg BID, or higher). Dose escalation follows a "3+3" design based on dose-limiting toxicity (DLT) assessment in the first 21-day cycle. Treatment continues until disease progression, unacceptable toxicity, or meeting other discontinuation criteria.
  Other Names: AZD3759, AZD9291

SUMMARY:
This is a clinical trial that aims to test Zorifertinib when used together with a known drug, Osimertinib. The goal is to learn if this combination is safe and works for people with advanced Non-Small Cell Lung Cancer (NSCLC) whose cancer has spread to the membranes surrounding the brain and spinal cord (a condition called leptomeningeal metastases) after being treated with Osimertinib.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients must meet all of the following criteria.

1. The patient or the guardian is required to understand and sign the informed consent form of this study.
2. During the screening period, subjects must have a previous histological or cytological diagnosis of NSCLC with a sensitising EGFR mutation (including L858R and/or Exon19Del).
3. Only patients who have developed meningeal progression after osimertinib treatment (at a standard dose of 80 mg QD; if the dose is 160 mg QD, it must be reduced to 80 mg QD for at least 1 week before receiving study treatment) (new-onset meningeal progression, or patients with existing meningeal progression that is poorly controlled using osimertinib combined with available conventional treatment [CNS symptoms not relieved or CSF cytology not turning negative], but the available conventional treatment must be washed out for at least 4 weeks) and have no extracranial progression are allowed to be enrolled.
4. Subjects with leptomeningeal metastases should have the positive results of cerebrospinal fluid (CSF) cytology. Subjects with negative CSF cytology but highly suspected of leptomeningeal metastases in combination with CSF biochemical test and brain or spinal cord MRI imaging examination are allowed to be enrolled into the study.
5. Subjects with meningeal progression and brain parenchyma progression are allowed to be enrolled.
6. Subjects must have at least one repeatedly evaluable, measurable target lesion (intracranial and/or extracranial) according to mRECIST 1.1 criteria or a repeatedly evaluable lesion according to RANO-LM criteria.
7. Subjects must be ≥ 18 years old before signing the informed consent form (ICF).
8. If there are neurological symptoms, the following conditions must be met: Able to take and swallow oral medication; No need to increase the hormone dose to enhance control of central nervous system symptoms for at least 1 week before study treatment. If a patient is taking hormone for the purpose of treating endocrine dysfunction or tumor-related symptoms (not central nervous system-related), the dose must be stable or reduced within 5 days before the study medication. Note: The hormone dose should be stable 5 days before the baseline brain MRI.
9. All toxicities related to anti-tumor therapy (including radiotherapy) must have resolved to ≤ Grade 1 (CTCAE 5.0, it is sufficient for neurotoxicity related to platinum treatment to resolve to ≤ Grade 2 [CTCAE]) before starting the study treatment. Patients with alopecia of any grade are allowed to be enrolled.
10. The screening period examination of patients must meet the followings:

    * Neutrophil count ≥ 1.5 x 109/L
    * Platelet ≥ 100 x 109/L
    * Hemoglobin ≥ 9 g/dL
    * Blood creatinine ≤ 1.5 x ULN, or creatinine clearance (Cockcroft-Gault formula) ≥ 50 mL/min
    * Total bilirubin ≤ 1.5 x ULN (for patients with Gilbert's syndrome or metastases to liver, ≤3 x ULN is acceptable)
    * Glutamic-oxaloacetic transferase ≤ 2 x ULN (for patients with metastases to liver, ≤ 3 x ULN is acceptable)
    * Glutamic-pyruvic transaminase ≤ 2 x ULN (for patients with metastases to liver, ≤ 3 x ULN is acceptable)
11. The estimated survival time of subjects is ≥ 6 weeks.
12. Karnofsky Performance Status (KPS) scale score ≥ 60.

Exclusion Criteria:

Patients must not enter the study if any of the following exclusion criteria is met:

1. Subjects who plan to receive brain radiotherapy or intrathecal injection during the period from signing ICF to study medication.
2. Radiotherapy history within 28 days before study drug administration is not allowed for enrollment, and palliative radiation to the skeleton occurring within 14 days before study drug administration is also not allowed for enrollment.
3. Subjects who have undergone major surgery (e.g. intrathoracic, intraperitoneal or pelvic surgery) within 4 weeks prior to the first dose of study treatment or who have not yet recovered from the side effects associated with such surgery are not allowed to be enrolled.
4. In addition to NSCLC, there are other malignant tumors, or a history of other malignant tumors within 5 years, except for the following cases: Complete resection of skin basal cell and squamous cell carcinoma and radical resection of any type of carcinoma in situ.
5. Suffering from clinically significant and uncontrollable cardiac disorder and/or heart-related events within 6 months, such as:

(1) Unstable angina within 6 months before the screening period; (2) Myocardial infarction within 6 months before the screening period; (3) Documented history of heart failure (NYHA Class III-IV) or left ventricular ejection fraction (LVEF) < 50%; (4) Uncontrollable hypertension: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg, with or without antihypertensive drug treatment; the drugs are allowed to be adjusted before the screening period; (5) Ventricular arrhythmia; (6) Supraventricular or sinus arrhythmias but difficult to control with drugs; (7) Arrhythmias that cannot be controlled by other drugs; (8) QTcF >470 ms (mean value of three readings corrected using the Fridericia formula) during the screening period.

(9) The patient has any factors that increase the risk of QTc prolongation or arrhythmic events, such as electrolyte disturbances, including: Grade 2 or higher hypokalemia according to CTCAE (electrolyte disturbances should be corrected to ≤Grade 1 according to CTCAE and documented before the first dose); heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death in a first-degree relative under the age of 40, or any concomitant medication known to prolong the QT interval and lead to torsades de pointes.

6. Suffering from gastrointestinal disorders or serious impairment of gastrointestinal function, which may significantly affect drug absorption (e.g. ulcerative diseases, uncontrollable nausea, or vomiting, diarrhea, or malabsorption syndrome).

7. Unable to discontinue the following medications before the start of the study drug and during the study according to the withdrawal period provided in Appendix 13.6 (see Appendix 13.6 for specific withdrawal periods):

1. Strong CYP3A4 inducers or inhibitors;
2. Drugs mainly metabolised by CYP3A4;
3. Drugs that may cause QT interval prolongation or torsade de pointe. 8. Patients with a previous or concurrent HIV infection are not allowed to enroll. Patients who are HCV antibody positive can be enrolled if HCV-RNA is undetectable (the lower limit of normal for HCV-RNA detection is based on the test values of each site) and there is no concurrent hepatitis B virus (HBV) infection. HBV-infected individuals are allowed to be enrolled if they meet the following criteria: 1) Patients with active hepatitis B must meet the following conditions: Antiviral treatment is given for at least 6 weeks before starting study treatment, HBV DNA must be <100 IU/mL, and ALT and AST levels must be <ULN; 2) Patients with resolved hepatitis B or chronic hepatitis B must meet the following criteria: Patients have received prophylactic antiviral treatment for at least 2-4 weeks before the start of study treatment, transaminases have been below ULN for >6 months, and HBV DNA is below 100 IU/mL (if in an inactive carrier state) 9. Women who are pregnant or lactating. Women of childbearing potential are required to use highly effective contraceptive methods during the dosing period and for 3 months after discontinuation of the drug. Fertile males must also use highly effective contraceptive methods during the dosing period and for 6 months after discontinuation of the drug.

A woman of child-bearing potential is defined as a non-postmenopausal woman who has experienced menarche and has not undergone sterilization (hysterectomy or bilateral salpingo-oophorectomy) or has no other causes of permanent infertility (such as Mullerian agenesis) determined by the investigator. Postmenopause is defined as amenorrhea ≥ 12 months without other biological or physiological reasons.

10. Due to existence of other serious, acute or chronic medical diseases (e.g. uncontrollable diabetes or psychic disorder or abnormal laboratory tests), the investigators judged that participating in the study treatment may bring more risks to the subjects or make it difficult to explain the study results.

11. Previously suffering from interstitial lung disease, including clinically significant radiation pneumonia (e.g. affecting daily life or requiring treatment intervention).

12. Subjects who have previously received treatment with zorifertinib drug product or drug substance.

13. A clear known history of allergy to the active ingredient or excipients of zorifertinib or to drugs with a chemical structure or class similar to zorifertinib.

14. Due to other combined diseases or other factors, investigators judged that participating in the clinical trial may bring greater risks to subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-04-23 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Determination of Recommended Dose Based on Incidence of Dose-Limiting Toxicities (DLTs) | During the first 21 days of continuous administration for each participant in the dose-escalation phase.
  A composite endpoint to determine the recommended dose of Zorifertinib in combination with Osimertinib. This is based on the occurrence of protocol-defined Dose-Limiting Toxicities (DLTs) within treatment. The Recommended Dose (RD) is the highest dose level at which the DLT rate is deemed acceptable by the Safety Review Committee (SRC) for further evaluation in the expansion cohort.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose until last dose (up to 12 months).
  Frequency, severity, and relationship to study treatment of all AEs and SAEs.
Objective Response Rate (ORR) for Leptomeningeal Metastases (per RANO-LM) | From first dose until disease progression or death from any cause, assessed up to 12 months.
  Proportion of participants with leptomeningeal disease achieving a Complete Response (CR) or Partial Response (PR) as assessed by the investigator according to RANO-LM neuroimaging criteria.
Leptomeningeal Progression-Free Survival (LM-PFS) (per RANO-LM) | From first dose until leptomeningeal progression or death from any cause, assessed up to 12 months.
  Time from first dose to the first documented progression in the leptomeninges according to RANO-LM criteria, or death from any cause, whichever occurs first
Leptomeningeal Progression-Free Survival (LM-PFS) Rate at 3, 6, and 9 Months | Assessed at 3, 6, and 9 months from first dose.
  Proportion of participants without leptomeningeal progression (as per RANO-LM criteria) at 3, 6, and 9 months after first dose.
Overall Survival (OS) Rate at 3, 6, and 9 Months | Assessed at 3, 6, and 9 months from first dose.
  Proportion of participants alive at 3, 6, and 9 months after first dose.
Cerebrospinal Fluid (CSF) Cytological Response Rate | CSF samples are collected at screening, at Week 6 (Day 22, corresponding to Cycle 2 Day 1 of a 21-day cycle), and every 6 weeks thereafter until disease progression, assessed up to 12 months.
  Proportion of participants achieving clearance of tumor cells (conversion from positive to negative cytology) in cerebrospinal fluid (CSF).
Complete Response (CR) Rate Based on Neurological Examination | Assessed at screening and at the end of every 21-day treatment cycle until disease progression, assessed up to 12 months.
  Proportion of participants achieving a Complete Response (CR) based on protocol-specified neurological examination.
Objective Response Rate (ORR) for Overall Tumors (per mRECIST 1.1) | From first dose until disease progression or death from any cause, assessed up to 12 months.
  Proportion of participants achieving Complete Response (CR) or Partial Response (PR) in overall systemic tumor burden, as assessed by the investigator using mRECIST 1.1 criteria.
Duration of Response (DoR) for Overall Tumors (per mRECIST 1.1) | From first documented response until progression or death, assessed up to 12 months.
  Time from the first documented overall tumor response (CR or PR) to the first documented overall disease progression or death due to any cause, whichever occurs first, assessed using mRECIST 1.1 criteria.
Progression-Free Survival (PFS) for Overall Tumors (per mRECIST 1.1) | From first dose until overall progression or death, assessed up to 12 months.
  Time from first dose to the first documented overall disease progression as per mRECIST 1.1 criteria, or death from any cause, whichever occurs first.
Objective Response Rate (ORR) for Intracranial Tumors (per mRECIST 1.1) | From first dose until intracranial disease progression or death from any cause, assessed up to 12 months.
  Proportion of participants achieving Complete Response (CR) or Partial Response (PR) in intracranial tumor burden, as assessed by the investigator using mRECIST 1.1 criteria.
Duration of Response (DoR) for Intracranial Tumors (per mRECIST 1.1) | From first documented response until intracranial progression or death, assessed up to 12 months.
  Time from the first documented intracranial tumor response (CR or PR) to the first documented intracranial disease progression or death due to any cause, whichever occurs first, assessed using mRECIST 1.1 criteria.
Change in Neurological Assessment in Neuro-Oncology (NANO) Score | Assessed at screening, on Days 1, 8, 15 (Cycle 1), and at the end of each subsequent 21-day treatment cycle until the End of Treatment visit, assessed up to 12 months.
  Change from baseline in the Neurological Assessment in Neuro-Oncology (NANO) score, as specified for leptomeningeal metastasis (NANO-LM). The NANO scale evaluates 9 neurological domains, with an overall response score where higher scores indicate worsening neurological function.
Progression-Free Survival (PFS) for Intracranial Tumors (per mRECIST 1.1) | From first dose until intracranial progression or death, assessed up to 12 months.
  Time from first dose to the first documented intracranial disease progression as per mRECIST 1.1 criteria, or death from any cause, whichever occurs first.

OTHER OUTCOMES:
Correlation of Biomarker Status in Cerebrospinal Fluid (CSF) with Clinical Efficacy | CSF samples for analysis are collected at Screening, at Week 6 (Cycle 2 Day 1 of a 21-day cycle), and at the time of suspected disease progression; efficacy outcomes are assessed throughout the study, up to 12 months.
  The correlation between the presence/level of specific biomarkers (e.g., genetic alterations) in cerebrospinal fluid (CSF) and clinical efficacy outcomes (e.g., objective response rate, progression-free survival).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou Q, Song Y, Zhang X, Chen GY, Zhong DS, Yu Z, Yu P, Zhang YP, Chen JH, Hu Y, Feng GS, Song X, Shi Q, Yang LL, Zhang PH, Wu YL. A multicenter survey of first-line treatment patterns and gene aberration test status of patients with unresectable Stage IIIB/IV nonsquamous non-small cell lung cancer in China (CTONG 1506). BMC Cancer. 2017 Jul 3;17(1):462. doi: 10.1186/s12885-017-3451-x. PMID 28673332
- [Result] Yin K, Li YS, Zheng MM, Jiang BY, Li WF, Yang JJ, Tu HY, Zhou Q, Zhong WZ, Yang XN, Chen HJ, Yan HH, Li LL, Wu YL, Zhang XC. A molecular graded prognostic assessment (molGPA) model specific for estimating survival in lung cancer patients with leptomeningeal metastases. Lung Cancer. 2019 May;131:134-138. doi: 10.1016/j.lungcan.2019.03.015. Epub 2019 Mar 18. PMID 31027690
- [Result] Yang JCH, Kim DW, Kim SW. Osimertinib activity in patients (pts) with leptomeningeal (LM) disease from non-small cell lung cancer (NSCLC): Updated results from BLOOM, a phase I study. [J]. Journal of Clinical Oncology, 2016, 34(15_suppl):9002-9002.
- [Result] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Result] Schag CC, Heinrich RL, Ganz PA. Karnofsky performance status revisited: reliability, validity, and guidelines. J Clin Oncol. 1984 Mar;2(3):187-93. doi: 10.1200/JCO.1984.2.3.187. PMID 6699671
- [Result] Omuro AM, Kris MG, Miller VA, Franceschi E, Shah N, Milton DT, Abrey LE. High incidence of disease recurrence in the brain and leptomeninges in patients with nonsmall cell lung carcinoma after response to gefitinib. Cancer. 2005 Jun 1;103(11):2344-8. doi: 10.1002/cncr.21033. PMID 15844174
- [Result] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Result] Le Rhun E, Weller M, Brandsma D, Van den Bent M, de Azambuja E, Henriksson R, Boulanger T, Peters S, Watts C, Wick W, Wesseling P, Ruda R, Preusser M; EANO Executive Board and ESMO Guidelines Committee. EANO-ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up of patients with leptomeningeal metastasis from solid tumours. Ann Oncol. 2017 Jul 1;28(suppl_4):iv84-iv99. doi: 10.1093/annonc/mdx221. No abstract available. PMID 28881917
- [Result] Janne PA, Yang JC, Kim DW, Planchard D, Ohe Y, Ramalingam SS, Ahn MJ, Kim SW, Su WC, Horn L, Haggstrom D, Felip E, Kim JH, Frewer P, Cantarini M, Brown KH, Dickinson PA, Ghiorghiu S, Ranson M. AZD9291 in EGFR inhibitor-resistant non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1689-99. doi: 10.1056/NEJMoa1411817. PMID 25923549
- [Result] Jackman DM, Holmes AJ, Lindeman N, Wen PY, Kesari S, Borras AM, Bailey C, de Jong F, Janne PA, Johnson BE. Response and resistance in a non-small-cell lung cancer patient with an epidermal growth factor receptor mutation and leptomeningeal metastases treated with high-dose gefitinib. J Clin Oncol. 2006 Sep 20;24(27):4517-20. doi: 10.1200/JCO.2006.06.6126. No abstract available. PMID 16983123
- [Result] Iuchi T, Shingyoji M, Itakura M, Yokoi S, Moriya Y, Tamura H, Yoshida Y, Ashinuma H, Kawasaki K, Hasegawa Y, Sakaida T, Iizasa T. Frequency of brain metastases in non-small-cell lung cancer, and their association with epidermal growth factor receptor mutations. Int J Clin Oncol. 2015 Aug;20(4):674-9. doi: 10.1007/s10147-014-0760-9. Epub 2014 Oct 22. PMID 25336382
- [Result] Gow CH, Chien CR, Chang YL, Chiu YH, Kuo SH, Shih JY, Chang YC, Yu CJ, Yang CH, Yang PC. Radiotherapy in lung adenocarcinoma with brain metastases: effects of activating epidermal growth factor receptor mutations on clinical response. Clin Cancer Res. 2008 Jan 1;14(1):162-8. doi: 10.1158/1078-0432.CCR-07-1468. PMID 18172267
- [Result] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- [Result] Eichler AF, Kahle KT, Wang DL, Joshi VA, Willers H, Engelman JA, Lynch TJ, Sequist LV. EGFR mutation status and survival after diagnosis of brain metastasis in nonsmall cell lung cancer. Neuro Oncol. 2010 Nov;12(11):1193-9. doi: 10.1093/neuonc/noq076. Epub 2010 Jul 13. PMID 20627894
- [Result] Liao BC, Lee JH, Lin CC, Chen YF, Chang CH, Ho CC, Shih JY, Yu CJ, Yang JC. Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors for Non-Small-Cell Lung Cancer Patients with Leptomeningeal Carcinomatosis. J Thorac Oncol. 2015 Dec;10(12):1754-61. doi: 10.1097/JTO.0000000000000669. PMID 26334749
- [Result] Ballard P, Yates JW, Yang Z, Kim DW, Yang JC, Cantarini M, Pickup K, Jordan A, Hickey M, Grist M, Box M, Johnstrom P, Varnas K, Malmquist J, Thress KS, Janne PA, Cross D. Preclinical Comparison of Osimertinib with Other EGFR-TKIs in EGFR-Mutant NSCLC Brain Metastases Models, and Early Evidence of Clinical Brain Metastases Activity. Clin Cancer Res. 2016 Oct 15;22(20):5130-5140. doi: 10.1158/1078-0432.CCR-16-0399. Epub 2016 Jul 19. PMID 27435396
- [Result] Armstrong TS，Mendoza T，Gning I，et al. Validation of the M. D. Anderson symptom inventory brain tumor module （MDASI-BT）［J］. J Neurooncol，2006，80（1）：27-35.
- [Result] Armstrong TS, Cohen MZ, Eriksen L, Cleeland C. Content validity of self-report measurement instruments: an illustration from the development of the Brain Tumor Module of the M.D. Anderson Symptom Inventory. Oncol Nurs Forum. 2005 May 10;32(3):669-76. doi: 10.1188/05.ONF.669-676. PMID 15897941
- [Result] Aparicio A, Chamberlain MC. Neoplastic meningitis. Curr Neurol Neurosci Rep. 2002 May;2(3):225-35. doi: 10.1007/s11910-002-0081-7. PMID 11937001
- [Result] Ahn MJ, Tsai CM, Shepherd FA, Bazhenova L, Sequist LV, Hida T, Yang JCH, Ramalingam SS, Mitsudomi T, Janne PA, Mann H, Cantarini M, Goss G. Osimertinib in patients with T790M mutation-positive, advanced non-small cell lung cancer: Long-term follow-up from a pooled analysis of 2 phase 2 studies. Cancer. 2019 Mar 15;125(6):892-901. doi: 10.1002/cncr.31891. Epub 2018 Dec 4. PMID 30512189
- [Result] Ahn MJ, Chiu CH, Cheng Y, Han JY, Goldberg SB, Greystoke A, Crawford J, Zhao Y, Huang X, Johnson M, Vishwanathan K, Yates JWT, Brown AP, Mendoza-Naranjo A, Mok T. Osimertinib for Patients With Leptomeningeal Metastases Associated With EGFR T790M-Positive Advanced NSCLC: The AURA Leptomeningeal Metastases Analysis. J Thorac Oncol. 2020 Apr;15(4):637-648. doi: 10.1016/j.jtho.2019.12.113. Epub 2019 Dec 27. PMID 31887431